CLINICAL TRIAL: NCT00455884
Title: International Cooperative Metabolic Study (iNCMS) of NutropinAq® [Somatropin (rDNA Origin) Injection] Replacement Therapy in Adults With Growth Hormone Deficiency
Brief Title: A Post Marketing Surveillance Study for NutropinAq® in Adults With Growth Hormone Deficiency
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: 2-79-58035-006
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Growth Hormone Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a multicenter, open-label, observational, post marketing surveillance program to collect information on the use of NutropinAq® in adults suffering from Growth Hormone Deficiency in Germany, Italy, and United Kingdom

ELIGIBILITY:
Inclusion Criteria:

* Patients with Growth Hormone Deficiency
* Patients treated with NutropinAq®
* Patients having completed growth (fused epiphyses)

Exclusion Criteria:

* Active neoplasia
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients treated with NutropinAq in the specialised adult endocrinology centres in Germany, Italy, and UK.
Sampling Method: Non-Probability Sample
Enrollment: 546 (Actual)
Dates: Start 2006-06; Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events | when reported

SECONDARY OUTCOMES:
Incidence of targeted adverse events, including adrenal insufficiency, arthritis, carpal tunnel syndrome, intracranial hypertension, new onset and recurrence of leukemia & tumor, pancreatitis, peripheral edema requiring medical intervention and death | when reported
Incidence of intercurrent cardiovascular events | when reported
Incidence of fractures | when reported

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Central Contact, Slough, Berkshire, United Kingdom